CLINICAL TRIAL: NCT05815303
Title: XELOX Combined With Cadonilimab Versus XELOX as Neoadjuvant Treatment for MRF-negative Locally Advanced, pMMR Rectal Cancer: a Randomised, Phase 2 Trial
Brief Title: XELOX Combined With Cadonilimab Versus XELOX as Neoadjuvant Treatment for Locally Advanced, pMMR Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, AIPING ZHOU, Vice director of Department of Medical Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC3627
Record Dates: First submitted 2023-04-01; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Rectal Cancer; MSS
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cadonilimab + XELOX (Experimental): Oxaliplatin 130 mg/m2 iv and Cadonilimab 10mg/kg iv on day 1； Capecitabine 1000mg/m2 po bid on day 1 to 14； every 21 day as a cycle, 4 cycles before surgery and 4 cycles after surgery
  Interventions: Drug: Cadonilimab; Drug: Oxaliplatin; Drug: Capecitabine
- XELOX (Sham Comparator): Oxaliplatin 130 mg/m2 iv on day 1； Capecitabine 1000mg/m2 po bid on day 1 to 14； every 21 day as a cycle, 4 cycles before surgery and 4 cycles after surgery
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Cadonilimab — 10mg/kg iv on day 1, every 21 day
  Arms: Cadonilimab + XELOX
Drug: Oxaliplatin — 130mg/m2 iv on day 1, every 21 day
Drug: Capecitabine — 1000mg/m2 po bid on day 1 to 14, every 21 day

SUMMARY:
This is a two-arm, open label, randomized phase II clinical study. The aim is to evaluate the safety and efficacy of Cadonilimab (a PD-1/CTLA-4 bispecific antibody) combined with XELOX regimen in pMMR locally advanced rectal cancer during the perioperative period. Eligible patients will receive either Cadonilimab plus XELOX or XELOX alone for 4 cycles before and 4 cycles after surgery. The primary endpoint is the pathological complete response rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or pathologically confirmed rectal adenocarcinoma located within 5 to 15cm from the anus with a stage of T3-4a or N+ according to the CT or endoscope
* Mesorectal fascia uninvolved
* Sign the informed consent form
* 18 years and older
* Mismatch repair proficient determined by immunohistochemistry
* No prior treatment
* Performance status: ECOG 0-1
* Good organ function:

Blood routine: hemoglobin ≥90g/L, neutrophil ≥1.5×10^9/L, platelet ≥100×10^9/L; Renal function: creatinine≤1.5×upper limit of normal (UNL) or creatinine clearance ≥50ml/min; Liver function: total bilirubin (TBIL)≤1.5×upper limit of normal (UNL); ALT≤2.5×UNL, AST≤2.5×UNL; Ejection fraction at least 50% (or lower limit of normal) by echocardiogram

Exclusion Criteria:

* Other pathological category, such as squamous cancer
* Distant metastasis or peritoneum implantation
* Have received chemotherapy or radiotherapy in the past
* Known to have allergic reactions to any ingredients or excipients of experimental drugs
* Unable to swallow or under other circumstance which would drug absorption
* Other active malignant tumors, excluding those who have been disease free for more than 5 years or in situ cancer considered to have been cured by adequate treatment
* Have received colorectal cancer surgery
* Diabetes was not controlled, defined as HbA1c > 7.5% after anti-diabetic drugs or hypertension was not controlled, defined as systolic / diastolic blood pressure > 140 / 90 mmHg after antihypertensive drug
* Myocardial infarction, severe/unstable angina, New York Heart Association (NYHA) class III or IV congestive heart failure in the past 12 months
* Known to be infected with human immunodeficiency virus (HIV), have acquired immunodeficiency syndrome (AIDS) related diseases, have active hepatitis B or hepatitis C
* Pregnant or nursing
* May increase the risk associated with participation in the study or administration of the study drug or mental illness that may interfere with the interpretation of research results
* There are other serious diseases that the researchers believe patients cannot be included in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
pCR | 3 years
  the rate of pathological complete response

SECONDARY OUTCOMES:
MPR | 3 years
  the rate of major pathological response according to Becker-TRG
DFS | From date of initiation of treatment to date of progression or death due to any cause, whichever occurs first, assessed up to 3 years
  disease free survival
OS | From date of initiation of treatment to date of death, assessed up to 3 years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided